CLINICAL TRIAL: NCT05933551
Title: Evaluation of the Efficiency of Training for Nurses to Use the Z Technique in Intramuscular Injection Application
Brief Title: Evaluation of the Efficiency of Z Technique Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nadiye BARIŞ EREN, Ass. Prof., Tarsus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TarsusU-NBARISEREN-001
Record Dates: First submitted 2023-06-26; First posted 2023-07-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2023-06

CONDITIONS: Nurse's Role
Keywords: Z technique; intramuscular enjection; skill; nurse; ventrogluteal region

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- After the training, the knowledge levels and skills of the nurses about the Z technique (Experimental)
  Interventions: Other: Z Technique Training

INTERVENTIONS:
Other: Z Technique Training — Training on Z technique will be given on the planned day, time and place. The education is planned to be given at Tarsus University. The training content will be presented to the participants as a powerpoint presentation (30 min), laboratory practice (15 min) and question-answer (15 min).

SUMMARY:
The goal of this clinical trial is to evaluate of the efficiency of training for nurses to use the Z technique in intramuscular injection application.

The main question it aims to answer is:

• Is there an effect of training on the use of Z technique in intramuscular injection practice of nurses?

The sample size was calculated as a minimum of 64 people. It consists of nurses who volunteered to participate in the study.

DETAILED DESCRIPTION:
The research was designed in a semi-experimental single group in the pretest-posttest order and will be carried out in four stages:

In the 1st Stage: The socio-demographic characteristics of the nurses and their knowledge levels about the Z technique will be evaluated before the training.

In the 2nd stage: Training will be given on the Z technique on the planned day, time and place. The education is planned to be given at Tarsus University. The training content will be presented to the participants as a powerpoint presentation (30 min), laboratory practice (15 min) and question-answer (15 min).

In the 3rd Stage: After the training, the knowledge levels and skills of the nurses regarding the Z technique will be evaluated.

In the 4th Stage: 1 month after the training, the use cases of the Z technique will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All nurses who volunteer, work in the hospital and perform injections will take part in the research as participants.

Exclusion Criteria:

* Participants who do not continue the study or who express that they want to leave and who do not apply injections in the clinic they work will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Knowledge levels for the Z technique | 10 min
  After the training, the knowledge levels of the nurses about the Z technique will be evaluated.
Skill levels for the Z technique | 10 min
  After the training, the skill levels of the nurses about the Z technique will be evaluated.
Frequency of Using the Z Technique | 1 month after the training.
  Z technique use cases will be evaluated 1 month after the training.

SECONDARY OUTCOMES:
Nurses' Descriptive Characteristics | 10 min
  The sociodemographic and working characteristics of the nurses before the training and the characteristics of the use of the Z technique in intramuscular injection will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Nadiye BARIS EREN, Principal Investigator — Tarsus University
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmaz D, Khorshid L, Dedeoglu Y. The Effect of the Z-Track Technique on Pain and Drug Leakage in Intramuscular Injections. Clin Nurse Spec. 2016 Nov/Dec;30(6):E7-E12. doi: 10.1097/NUR.0000000000000245. PMID 27753676
- [Background] Altun I. May the Z-Tracking Technique to Prevent Any Leakage in Insulin Injection Be an Alternative to the 10-Second Waiting Technique? J Diabetes Sci Technol. 2018 Mar;12(2):537-538. doi: 10.1177/1932296817730378. Epub 2017 Sep 18. No abstract available. PMID 28918650
- [Background] Ayinde O, Hayward RS, Ross JDC. The effect of intramuscular injection technique on injection associated pain; a systematic review and meta-analysis. PLoS One. 2021 May 3;16(5):e0250883. doi: 10.1371/journal.pone.0250883. eCollection 2021. PMID 33939726
- See also: The Effect of Different Techniques Used in Intramuscular Injection On Pain And Drug Leakage — https://dergipark.org.tr/en/pub/iaaojh/issue/64539/773721